CLINICAL TRIAL: NCT04333108
Title: Phase 3 Study to Compare Oral Masitinib to Placebo in Treatment of Patients With Smouldering or Indolent Severe Systemic Mastocytosis, Unresponsive to Optimal Symptomatic Treatment
Brief Title: Masitinib in Severe Indolent or Smoldering Systemic Mastocytosis Unresponsive to Optimal Symptomatic Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB15003; 2016-001447-39 (EudraCT Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: Mastocytosis with handicap; Mastocytosis; Mast cell; Mast cell infiltration; Skin; Bone marrow; Pruritus; Flushes; c-kit; c-kit mutation; Wild Type; Mutation Asp-816-Val(D816V); Indolent systemic mastocytosis; smoldering systemic mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis; Pruritus; Blushing; Piebaldism | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib & BSC (Experimental): Experimental Arm:
  Masitinib (titration to 6.0 mg/kg/day) administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC).
  Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment, followed by dose escalation to 6.0 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control.
  Interventions: Drug: Masitinib; Other: Best Supportive Care
- Placebo & BSC (Placebo Comparator): Placebo Comparator:
  Matching placebo administered as an add-on to optimal concomitant symptomatic treatment (i.e. best supportive care, BSC)
  Interventions: Other: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: Masitinib — Masitinib 6 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib & BSC
Other: Placebo — Matching placebo
  Arms: Placebo & BSC
Other: Best Supportive Care — Optimal concomitant symptomatic treatments. Includes: H1- and H2-antihistamines, proton pump inhibitors (PPI), sodium cromoglycate, antidepressants, leukotriene antagonists and corticosteroids.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of oral masitinib versus placebo in the treatment of patients suffering from smouldering or indolent systemic mastocytosis with severe symptoms of mast cell mediator release, unresponsive to optimal symptomatic treatment.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor that modulates mast cell activity via inhibition of c-Kit, Lyn and Fyn kinase signaling pathways. This is a multicenter, randomized, double-blind, placebo-controlled, 2-parallel-group, trial comparing oral masitinib versus placebo in the treatment of patients suffering from smouldering or indolent systemic mastocytosis with severe symptoms of mast cell mediator release (also referred to as handicaps), unresponsive to optimal symptomatic treatment. The treatment period is 24 weeks. Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment, followed by dose escalation to 6.0 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with one of the following documented mastocytosis subtypes (variants): Smouldering Systemic Mastocytosis, Indolent Systemic Mastocytosis
2. An excess of mast cells or a presence of abnormal mast cells in at least two organs (among skin, bone-marrow and GI Tract).
3. Patient with documented systemic mastocytosis and evaluable disease based upon histological criteria
4. Patient with documented treatment failure of his/her symptom(s) (within the past 2 years) with at least two of the symptomatic treatments used at optimized dose: Anti H1, Anti H2, Proton pump inhibitor, Antidepressants, Cromoglycate Sodium, Antileukotriene.
5. Patient with severe symptoms of mastocytosis over the 14-day run-in period including at least one among pruritus, flushes, and depression: pruritus score ≥ 9, number of flushes per week ≥ 8, Hamilton rating scale for depression (HAMD-17) score ≥ 19.

Exclusion Criteria:

1. Patient with one of the following mastocytosis: Cutaneous Mastocytosis, Systemic Mastocytosis with an Associated clonal Hematologic Non Mast cell lineage Disease (SM-AHNMD), Mast cell leukemia (MCL), Aggressive systemic mastocytosis (ASM)
2. Previous treatment with any Tyrosine Kinase Inhibitor
3. Treatment with any investigational agent within 8 weeks prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative response (3R75%) | 24 weeks
  Cumulative response in at least one of three severe baseline symptoms of mast cell mediator release (pruritus, flushes, or depression). Response was defined as a 75% improvement from baseline for any of these three symptoms. Cumulative response was defined as the number of actual responses between weeks 8 and 24, divided by the total number of possible responses over the same treatment period (ie, with five scheduled visits, each patient had a maximum of five to 15 possible responses depending on the number of severe baseline symptoms).

SECONDARY OUTCOMES:
Cumulative response (4R75%) | 24 weeks
  Cumulative response in at least one of four severe baseline symptoms of mast cell mediator release (pruritus, flushes, depression, or asthenia). Response is defined as a 75% improvement from baseline for any of these four symptoms. Cumulative response was defined as the number of actual responses between weeks 8 and 24, divided by the total number of possible responses over the same treatment period (ie, with five scheduled visits, each patient had a maximum of five to 20 possible responses depending on the number of severe baseline symptoms).
Cumulative response (2R75%) | 24 weeks
  Cumulative response in at least one of two severe baseline symptoms of mast cell mediator release (pruritus or flushes). Response is defined as a 75% improvement from baseline for either of these two symptoms. Cumulative response is defined as the number of actual responses between weeks 8 and 24, divided by the total number of possible responses over the same treatment period (ie, with five scheduled visits, each patient had a maximum of five to 10 possible responses depending on the number of severe baseline symptoms).
Cumulative response | 24 weeks
  Cumulative response on each of the individual handicaps. Response is defined as a 75% improvement from baseline for either of these two symptoms. Cumulative response is defined as the number of actual responses between weeks 8 and 24, divided by the total number of possible responses over the same treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Bulai Livideanu, MD, MSc, Principal Investigator — Centre Hospitalier Universitaire, Service de Dermatologie, Toulouse -France
Locations (17):
- France (8):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hospital Jean-Minjoz, Besançon
  - Grenoble University Hospital, Grenoble
  - Hospital Claude Huriez, Lille
  - Marseille University Hospital Timone, Marseille
  - Centre de référence de Mastocytose (CEREMAST), Paris
  - Poitiers University Hospital, Poitiers
  - Centre Hospitalier Universitaire, Toulouse
- University Hospital Charité, Berlin, Germany
- Erasmus University Medical Center, Rotterdam, Netherlands
- Poland (2):
  - Medical University of Gdańsk, Gdansk
  - The University Hospital in Krakow (Szpital Uniwersytecki w Krakowie), Krakow
- University Hospital in Bucharest (Spitalul Universitar de Urgență București), Bucharest, Romania
- Almazov National Medical Research Centre, Saint Petersburg, Russia
- Ukraine (2):
  - Dnipropetrovsk Clinical Association of Emergency Medical Care of Dnipropetrovsk Regional, Dnipro
  - Private Enterprise Private Manufacturing Company Acinus, Poltava
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul C, Sans B, Suarez F, Casassus P, Barete S, Lanternier F, Grandpeix-Guyodo C, Dubreuil P, Palmerini F, Mansfield CD, Gineste P, Moussy A, Hermine O, Lortholary O. Masitinib for the treatment of systemic and cutaneous mastocytosis with handicap: a phase 2a study. Am J Hematol. 2010 Dec;85(12):921-5. doi: 10.1002/ajh.21894. PMID 21108325
- [Background] Lortholary O, Chandesris MO, Bulai Livideanu C, Paul C, Guillet G, Jassem E, Niedoszytko M, Barete S, Verstovsek S, Grattan C, Damaj G, Canioni D, Fraitag S, Lhermitte L, Georgin Lavialle S, Frenzel L, Afrin LB, Hanssens K, Agopian J, Gaillard R, Kinet JP, Auclair C, Mansfield C, Moussy A, Dubreuil P, Hermine O. Masitinib for treatment of severely symptomatic indolent systemic mastocytosis: a randomised, placebo-controlled, phase 3 study. Lancet. 2017 Feb 11;389(10069):612-620. doi: 10.1016/S0140-6736(16)31403-9. Epub 2017 Jan 7. PMID 28069279
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877